CLINICAL TRIAL: NCT03957213
Title: Enhancing Cognition in Older Adults With Intermittent Hypoxia and Cognitive Training: The EXCITE Study
Brief Title: Enhancing Cognition in Older Adults With Intermittent Hypoxia and Cognitive Training
Acronym: EXCITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: IRB201802556
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Aging
Keywords: Intermittent Hypoxia; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active IH + CT (Experimental): Acute intermittent hypoxia will be provided to the subject by delivering 15 brief exposures (~60 seconds) of hypoxic air alternated with 15 brief exposures (~60 seconds) of room air. The amount of oxygen delivered during hypoxic exposures may range from 15%-9% fraction of inspired oxygen, compared to 21% oxygen in normal atmospheric air. This is followed by a 30 minute rest period and then 60 minutes of computerized cognitive training.
  Interventions: Device: Acute Intermittent Hypoxia; Behavioral: Computerized Cognitive Training
- Sham IH + CT (Sham Comparator): A sham protocol will be administered in which 21% fraction of inspired oxygen will be delivered by the hypoxicator during hypoxic intervals, and room air will be delivered through the four-way valve during room air intervals. This is followed by a 30 minute rest period and then 60 minutes of computerized cognitive training (Posit; Brain HQ).
  Interventions: Behavioral: Computerized Cognitive Training

INTERVENTIONS:
Device: Acute Intermittent Hypoxia — Acute intermittent hypoxia is a safe, non-invasive technique. All sessions will be monitored by research study staff trained in delivering acute intermittent hypoxia. Hypoxic intervals will be delivered with a commercially available sports performance hypoxicator. A unit capable of delivering a fraction of inspired oxygen ranging from 21%-9% will be used. Air will be delivered into a mask that will be secured comfortably over the subject's nose and mouth. Intervention sessions will occur for 10 days over a 2 week period.
  Arms: Active IH + CT
Behavioral: Computerized Cognitive Training — 60 minutes of Double Decision cognitive training for 10 days over a 2 week period.

SUMMARY:
The current study will investigate methods for enhancing cognitive training (CT) effects in healthy older adults by employing a combination of interventions facilitating neural plasticity and optimizing readiness for learning. Adults over the age of 65 represent the fastest growing group in the US population. As such, age-related cognitive decline represents a major concern for public health. Recent research suggests that cognitive training in older adults can improve cognitive performance, with effects lasting up to 10 years. However, these effects are typically limited to the tasks trained, with little transfer to other cognitive abilities or everyday skills. A pilot randomized clinical trial will examine the individual and combined impact of pairing cognitive training with an intermittent hypoxia (IH) intervention. The investigators will compare changes in cognitive and brain function resulting from CT combined with active IH versus CT combined with sham IH using a comprehensive neurocognitive, clinical, and multimodal neuroimaging assessment of brain structure, function, and metabolic state. Functional magnetic resonance imaging (FMRI) will be used to assess brain response during speed of processing; the active cognitive abilities trained by CT. Magnetic resonance spectroscopy (MRS) will assess cerebral metabolites, including ATP and GABA concentrations sensitive to neural plasticity.

DETAILED DESCRIPTION:
Age-related cognitive decline has become a major public health concern. As the population ages, the number of older adults experiencing cognitive and functional disturbances has increased. There is currently a paucity of effective interventions to prevent or treat cognitive decline or to enhance brain function in the elderly. The proposed study will recruit a cohort from the state with the highest growth of older adults. The study team will employ a randomized controlled trial (RCT) to test whether the benefits of cognitive training (CT) can be enhanced by a combined adjunctive intervention aimed at increasing neural plasticity and optimizing readiness for learning: intermittent hypoxia (IH).

Current CT approaches have been shown to improve performance on trained tasks, with effects lasting up to ten years. However, generalization of effects to other cognitive domains and everyday functioning has been a problem in the past. There is now compelling evidence that the elderly do experience functional improvements that persist long after initial training, though peoples' ability to derive such benefits varies. Combined interventions have rarely been examined and methods aimed at increasing neural plasticity and optimizing readiness for learning are only now beginning to be explored. The proposed study will test one theoretical approach for facilitating and optimizing CT effects on functional outcome. The investigators will use an adjunctive physiological method to further stimulate task-related brain regions, directly enhancing neural responsivity/plasticity and ultimately learning. While theoretical rationales exist for each of these approaches, no studies to date have shown whether adjunctive administration can optimize learning and functional status in the elderly.

A pilot randomized clinical trial will enroll 55 participants, with a target of 20 participants completing the study, and as many as 30 participants consenting but failing to meet inclusion criteria at in person screening, and 5 participants withdrawing prior to completion. Cognitively healthy elderly adults, age 65-89 will undergo either a CT intervention in combination with IH or sham IH control. The CT intervention will employ the Double Decision task from the POSIT Science Brain HQ; a well validated CT method for enhancing cognitive functioning in the elderly. Participants will receive IH or sham/placebo IH administered during training.

Participants will be assessed at baseline and after CT (2 weeks). At each time point, a comprehensive neurocognitive, clinical and multimodal neuroimaging assessment of brain function, metabolic state, and brain structure will be conducted.

FMRI will be used to assess brain response during working memory, attention and memory encoding. Proton magnetic resonance spectroscopy (MRS) will assess cerebral metabolites, including gamma-aminobutyric acid (GABA) concentrations, sensitive to neural plasticity in task-associated brain regions.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Physically mobile
* Cognitive function between 0-79th percentile determined by screening results on the POSIT Baseline Cognitive Training computerized tasks.

Exclusion Criteria:

* Neurological disorders (e.g., dementia, stroke, seizures, traumatic brain injury).
* Evidence of dementia (NACC UDS scores of 1.5 standard deviations below the mean for age, sex and education adjusted norms in a single cognitive domain on the task).
* Past opportunistic brain infection
* Major psychiatric illness (schizophrenia, intractable affective disorder, current substance dependence diagnosis or severe major depression and/or suicidality.
* Unstable (e.g., cancer other than basal cell skin) and chronic (e.g, severe diabetes) medical conditions.
* MRI contraindications (e.g., pregnancy, claustrophobia, metal implants that are contraindicated for MRI).
* Physical impairment precluding motor response or lying still for 1 hr and inability to walk two blocks without stopping.
* Certain prescription CNS acting medications that alter the neuroplastic response of brain tissue (gabaergic and glutamatergic drugs).
* Hearing or vision deficits that will not allow for standardized cognitive training; ie colorblindness, inability to hear through headphones (with or without hearing aids), macular degeneration or other significant diseases that cause severe loss of vision. If vision is corrected with lenses to appropriate levels, then participant will be eligible.
* Left handedness, as those with left-handedness have a higher percentage rate of atypical functional lateralization for brain functions, which would significantly interfere with interpretability of brain data.
* Cancer (other than skin) within the last 3 years.
* Sleep apnea diagnosis or suspected sleep apnea.
* Heart failure or heart disease.
* Pulmonary disease.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Change in Posit Science Double Decision Performance | Baseline; Week 2
  Determine whether training performance improves when cognitive training (CT) is coupled with intermittent hypoxia (IH). Posit Science Double Decision is designed to improve the speed and accuracy with which the brain can process visual information, both at the center of gaze and on the periphery, known as "useful field of view" (UFOV). Scored in milliseconds, where lower scores indicate better processing speeds. CT will involve up to 10 hours of training over 2-weeks (10 days) and employs a PositScience BrainHQ suite via its researcher portal

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Woods, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No